CLINICAL TRIAL: NCT05536583
Title: Shanghai Tenth People's Hospital，School of Medicine, Tongji University
Brief Title: Clinical Efficacy and Safety of Laparoscopic Sleeve Gastrectomy in Obese Patients With PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSG in PCOS patients
Record Dates: First submitted 2022-09-06; First posted 2022-09-13 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; Laparoscopic sleeve gastrectomy; Obesity; menstrual cycle
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity

STUDY DESIGN:
Intervention Model Description: Comparison of obese patients with PCOS and simple obesity after laparoscopic sleeve gastrectomy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOS group (Experimental): Obese Patients with PCOS underwent LSG
  Interventions: Procedure: Laparoscopic sleeve Gastrectomy
- Control group (Active Comparator): Sample obese patients without PCOS underwent LSG
  Interventions: Procedure: Laparoscopic sleeve Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve Gastrectomy — Laparoscopic sleeve Gastrectomy

SUMMARY:
This study aims to evaluate the clinical efficacy and safety in obese patients with Polycystic Ovary Syndrome after laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical efficacy and safety of laparoscopic sleeve gastrectomy in obese patients with Polycystic Ovary Syndrome（PCOS). About 100 obese patients with PCOS and 100 simple obese patients (without complications) were enrolled.

All PCOS patients with obesity underwent LSG. A multidisciplinary team evaluated participants with obesity at baseline, 1, 3, 6, 12, 24, and 36 months after LSG. Anthropometrics, Metabolic indicators, sex hormones, menstruation，glucose-lipid metabolic markers, and hepatic steatosis were measured baseline and postoperative.

ELIGIBILITY:
Inclusion Criteria:

* age ranged from 18~45 years old,
* BMI over 37.5 kg/m2, or BMI over 32.5 kg/m2 with diabetes which meets the recommended cutoff for bariatric surgery of the Guidelines for surgical treatment of obesity accompanied with or without type 2 diabetes in China.

Exclusion Criteria:

* outside of the 18-45 age range;
* secondary obesity caused by endocrine disorders;
* history of more than one bariatric procedure;
* severe hepatic, renal or heart dysfunction;
* mental illnesses or intellectual disability.
* pregnancy or lactation
* contraindications for laparoscopic surgery, such as gastrointestinal diseases of intra-abdominal infection, adhesions, etc.,

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Menstrual cycles | 3 years
  the total number of menstrual periods in the last year

SECONDARY OUTCOMES:
ZAG | 3 years
  zinc-alpha2-glycoprotein
FGF-19 | 3 years
  fibroblast growth factor 19
FGL-1 | 3 years
  fibrinogen-like protein 1
BMI | 3 years
  BMI=weight(kg)/height(m)^2
Waist/hip Ratio | 3 years
  WHR=Waist Circumference in centimeter/Hip Circumference in centimeter
TT | 3 years
  total testosterone in nmol/L
FBG | 3 years
  fasting blood-glucose in mmol/L
PBG | 3 years
  postprandial blood-glucose in mmol/L
FINS | 3 years
  fasting serum insulin in mU/L
PINS | 3 years
  postprandial insulin in mU/L
ALT | 3 years
  alanine aminotransferase in U/L
AST | 3 years
  aspartate aminotransferase in U/L
UA | 3 years
  Uric acid in umol/L
HOMA-IR | 3 years
  Homeostatic model assessment insulin resistance index=FBG*FINS/22.5
HbA1c (%) | 3 years
  Glycated hemoglobin
SHBG | 3 years
  sex hormone-binding globulin in nmol/L
FT | 3 years
  free testosterone (nmol/L)
DHEAS | 3 years
  Dehydroepiandrosterone Sulfate (ug/dl)
LDL-C | 3 years
  low-density lipoprotein cholesterol in mmol/L
HDL-C | 3 years
  Hight-density lipoprotein cholesterol in mmol/L
Fertility | 3 years
  sexual function, fertility
LH | 3 years
  luteinizing hormone in IU/L
FSH | 3 years
  follicle-stimulating hormone in IU/l
E2 | 3 years
  Estradiol in pmol/L
PRL | 3 years
  Prolactin in uIU/ml
CR | 3 years
  Creatinine in umol/L
AD | 3 years
  Androstenedione in ng/ml
TC | 3 years
  Total Cholesterol (mmol/L)
TG | 3 years
  Triglyceride (mmol/L)